CLINICAL TRIAL: NCT05152225
Title: Neurological Complication of Infective Endocarditis: A Prospective Multi-site Cohort Study With Systematic MRI and Digital Subtraction Angiography
Brief Title: Neurological Complication of Infective Endocarditis: A Prospective Multi-site Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: the Jeunes en Neuroradiologie Interventionnelle (JENI) research group (Network)
Collaborators: University Hospital, Limoges (Other); Sainte Anne Hospital (Paris) (Unknown)
Responsible Party: Principal Investigator, Basile Kerleroux, MD-MSc, the Jeunes en Neuroradiologie Interventionnelle (JENI) research group
Other Study IDs: JENI2021IIA
Record Dates: First submitted 2021-11-24; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Endocarditis, Bacterial; Aneurysm, Intracranial Mycotic
Keywords: MRI; digital subtraction angiography
MeSH Terms: conditions — Endocarditis, Bacterial; Intracranial Aneurysm | interventions — Angiography, Digital Subtraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infective endocarditis: Infective endocarditis with systematic brain MRI and digital subtraction angiography (DSA) performed routinely.
  Interventions: Diagnostic Test: Brain MRI; Diagnostic Test: digital subtraction angiography (DSA)

INTERVENTIONS:
Diagnostic Test: Brain MRI — Brain MRI performed routinely in patients with EI
Diagnostic Test: digital subtraction angiography (DSA) — Digital Subtraction Angiography (DSA) performed routinely in patients with EI

SUMMARY:
The main objective of this study is to better estimate the rate of infectious intracranial aneurysms (IIA) in proved infective endocarditis (IE). It also aims to identify MRI markers capable of accurately predicting (or excluding) IIA; to assess the impact of the different MRI abnormalities on the outcome; to capture the real-world management of EI with neurological complications in comprehensive IE centers in France

DETAILED DESCRIPTION:
Rationale:

The incidence of Infective endocarditis (IE) in developed countries is approximately 3-15 per 100,000 pers-years. Discharge mortality remains 15-30% and therapeutic management suffers in many ways from the paucity of randomized studies.(1) Symptomatic neurological complications, which occur in 15 to 30% of patients, are the most frequent extra-cardiac complication of IE and are deemed to worsen the outcome of EI.(2,3) Among this overall neurological complications, Infectious Intracranial Aneurysms (IIA) are a relatively rare, yet probably underestimate, vessel wall injury caused by septic emboli, with potentially intracranial bleeding for the patients.

Neuroimaging in the context of IE has gained wide acceptance and is encouraged in the current guidelines.(4,5) Nevertheless the benefit of early neuroimaging to optimize the initial therapeutic management remains debated.(6,7) While the appearance and the frequency of the various neurologic complications of EI are well known thanks to prospective cohort studies with systematic pre-therapeutic MRI(8-10), several clinically relevant questions are still unknow or approximate, including: 1/ What is the rate of IIA in proved EI. The current gold standard for the detection of these small and distally located aneurysms remains Digital Subtraction Angiography (DSA) and to our knowledge, there is no prospective unbiased cohort of IE with systematic DSA available in the literature. 2/ Are there MRI signs correlated with the presence of IIA on DSA? Several MRI markers such as sulcal SWI lesion or cerebral microbleeds (CMBs) with contrast enhancement look promising (10), but validation in unbiased prospective studies with systematic MRI and DSA is needed. 3/ What is the impact on the outcome of the different MRI abnormalities and of unruptured and ruptured IIA? As previously mentioned, the value of both MRI and DSA remain unclear to guide the acute therapeutic management of EI. A recent French survey highlighted differences between university Hospital in France in the management of IIA. Thus, the analysis of the current management of EI with neurological complications could also help at informing the design of future randomized trials.

Questions:

1. Better estimate the rate of IIA in proved EI.
2. Identify MRI markers able to accurately predict (or exclude) IIA.
3. What is the impact of different MRI abnormalities on the outcome?
4. Capture the real-world management of EI with neurological complications in comprehensive EI centers in France

Design and setting:

Multi-site, prospective cohort study, with standardized imaging protocol, in academic centers where MRI and DSA are performed routinely in patients with EI.

Ethics:

As for all non-interventional studies of de-identified data, written informed consent will be waived and a commitment to compliance (Reference Methodology CPMR-4) will be filed to the French data protection authority (CNIL) prior to data centralization, in respect to the General Data Protection Regulation. Patients and proxies will be informed they could oppose the use of their data for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* patients with left-sided active infective endocarditis (IE) satisfying modified Duke Criteria,
* patients who underwent both digital subtraction angiography (DSA) and brainMRI (as part of routine care)
* DSA protocol with 3D rotational for both carotids and one vertebral artery
* MRI/MRA standardized protocol including at least: Diffusion, FLAIR, 3D SWI, 3DT1SE and post gadolinium 3DT1SE and 3D TOF (large field: from the vertex to the magnum foramen).

Exclusion Criteria:

* uncertain diagnosis of IE by infectious disease consultants
* patients with chronic IE
* MRI performed after the completion of Infectious intracranial aneurysms (IIA) treatment
* MRI performed without contrast injection or complete protocol
* More than 48-hours delay between performing MRI and DSA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter, prospective cohort study of infective endocarditis in academic centers where Brain MRI and DSA are performed routinely.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The assess the occurrence of infectious intracranial aneurysms in proven infective endocarditis | 3 months
  In all included cases, infectious intracranial aneurysms will be detected using cerebral Digital Subtraction Angiography (DSA), which remains the current gold standard for the detection of these small and distally located aneurysms. DSA protocol will include 2D and 3D rotational acquisitions on both carotid arteries and one vertebral artery. The number of infective endocarditis with infectious intracranial aneurysms will be referred to the total number of endocarditis to estimate the incidence of these cerebral anomalies.

SECONDARY OUTCOMES:
To assess the diagnostic performance of MRI markers to detect infectious intracranial aneurysms | 3 months
  Logistic regression and Linear Discriminant Analysis (LDA) methods will be used to identify the most relevant MRI signs to predict or exclude IIA (on DSA).
To assess the predictive performance of imaging markers on clinical outcome | 2 years
  Logistic regression will be used to identify MRI and DSA sign associated with neurological worsening at follow-up.
To assess the rate of symptomatic intracranial haemorrhage following heart surgery | 6 months
  In case of neurological deterioration after cardiac surgery, brain imaging (MRI or NCCT) will be performed to detect the occurrence or progression of cerebral haemorrhage. Logistic regression will be used to identify the MRI and DSA signs associated with this neurological complication.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carneiro TS, Awtry E, Dobrilovic N, Fagan MA, Kimmel S, Weinstein ZM, Cervantes-Arslanian AM. Neurological Complications of Endocarditis: A Multidisciplinary Review with Focus on Surgical Decision Making. Semin Neurol. 2019 Aug;39(4):495-506. doi: 10.1055/s-0039-1688826. Epub 2019 Sep 18. PMID 31533190
- [Result] Garcia-Cabrera E, Fernandez-Hidalgo N, Almirante B, Ivanova-Georgieva R, Noureddine M, Plata A, Lomas JM, Galvez-Acebal J, Hidalgo-Tenorio C, Ruiz-Morales J, Martinez-Marcos FJ, Reguera JM, de la Torre-Lima J, de Alarcon Gonzalez A; Group for the Study of Cardiovascular Infections of the Andalusian Society of Infectious Diseases; Spanish Network for Research in Infectious Diseases. Neurological complications of infective endocarditis: risk factors, outcome, and impact of cardiac surgery: a multicenter observational study. Circulation. 2013 Jun 11;127(23):2272-84. doi: 10.1161/CIRCULATIONAHA.112.000813. Epub 2013 May 6. PMID 23648777
- [Result] Snygg-Martin U, Gustafsson L, Rosengren L, Alsio A, Ackerholm P, Andersson R, Olaison L. Cerebrovascular complications in patients with left-sided infective endocarditis are common: a prospective study using magnetic resonance imaging and neurochemical brain damage markers. Clin Infect Dis. 2008 Jul 1;47(1):23-30. doi: 10.1086/588663. PMID 18491965
- [Result] Baddour LM, Wilson WR, Bayer AS, Fowler VG Jr, Tleyjeh IM, Rybak MJ, Barsic B, Lockhart PB, Gewitz MH, Levison ME, Bolger AF, Steckelberg JM, Baltimore RS, Fink AM, O'Gara P, Taubert KA; American Heart Association Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease of the Council on Cardiovascular Disease in the Young, Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and Stroke Council. Infective Endocarditis in Adults: Diagnosis, Antimicrobial Therapy, and Management of Complications: A Scientific Statement for Healthcare Professionals From the American Heart Association. Circulation. 2015 Oct 13;132(15):1435-86. doi: 10.1161/CIR.0000000000000296. Epub 2015 Sep 15. PMID 26373316
- [Result] Habib G, Lancellotti P, Antunes MJ, Bongiorni MG, Casalta JP, Del Zotti F, Dulgheru R, El Khoury G, Erba PA, Iung B, Miro JM, Mulder BJ, Plonska-Gosciniak E, Price S, Roos-Hesselink J, Snygg-Martin U, Thuny F, Tornos Mas P, Vilacosta I, Zamorano JL; ESC Scientific Document Group. 2015 ESC Guidelines for the management of infective endocarditis: The Task Force for the Management of Infective Endocarditis of the European Society of Cardiology (ESC). Endorsed by: European Association for Cardio-Thoracic Surgery (EACTS), the European Association of Nuclear Medicine (EANM). Eur Heart J. 2015 Nov 21;36(44):3075-3128. doi: 10.1093/eurheartj/ehv319. Epub 2015 Aug 29. No abstract available. PMID 26320109
- [Result] Iung B, Tubiana S, Klein I, Messika-Zeitoun D, Brochet E, Lepage L, Al-Attar N, Ruimy R, Leport C, Wolff M, Duval X; ECHO-IMAGE Study Group. Determinants of cerebral lesions in endocarditis on systematic cerebral magnetic resonance imaging: a prospective study. Stroke. 2013 Nov;44(11):3056-62. doi: 10.1161/STROKEAHA.113.001470. Epub 2013 Sep 3. PMID 24003046
- [Result] Cho SM, Rice C, Marquardt RJ, Zhang LQ, Khoury J, Thatikunta P, Buletko AB, Hardman J, Uchino K, Wisco D; Infective Endocarditis Strokes and Imaging Characteristics (IESIC) group. Magnetic Resonance Imaging Susceptibility-Weighted Imaging Lesion and Contrast Enhancement May Represent Infectious Intracranial Aneurysm in Infective Endocarditis. Cerebrovasc Dis. 2017;44(3-4):210-216. doi: 10.1159/000479706. Epub 2017 Aug 19. PMID 28848178
- [Result] Migdady I, Rice CJ, Hassett C, Zhang LQ, Wisco D, Uchino K, Cho SM. MRI Presentation of Infectious Intracranial Aneurysms in Infective Endocarditis. Neurocrit Care. 2019 Jun;30(3):658-665. doi: 10.1007/s12028-018-0654-1. PMID 30519794